CLINICAL TRIAL: NCT06297785
Title: Online, Gut-directed Hypnotherapy for Patients With Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Simrén, Professor, MD, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-03997-01
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: IBS - Irritable Bowel Syndrome
Keywords: Gut-directed hypnotherapy
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nurse-delivered, gut-directed hypnotherapy (Other)
  Interventions: Behavioral: Gut-directed hypnotherapy

INTERVENTIONS:
Behavioral: Gut-directed hypnotherapy — Gut-directed hypnotherapy for patients with irritable bowel syndrome (IBS). Gut-directed hypnotherapy (8 sessions), will be given online in a group setting.The hypnosis treatment is administered by a nurse specially trained in Cognitive Behavioral Therapy (CBT) and hypnotherapy. The treatment is based on the North Carolina protocol. Patients will assess gastro-intestinal symptom severity before, during and after treatment, as well as at follow-up.

SUMMARY:
Adult IBS patients with symptoms refractory to standard medical treatment will receive online nurse-administered, gut-directed hypnotherapy in groups. The primary outcome measure was change in gastro-intestinal symptom severity. Secondary outcomes are GI-specific anxiety, general anxiety and depression, quality of life, and extracolonic symptom severity. Usability of the digital platform as well as patient treatment satisfaction will also be assessed.

DETAILED DESCRIPTION:
IBS patients with symptoms refractory to standard treatment and who were referred to a specialist unit for hypnotherapy, will be included in the study consecutively. The patients will receive gut-directed hypnotherapy given by a nurse trained in Cognitive Behavioral Therapy (CBT) and hypnotherapy. Effects of treatment will be measured by validated questionnaires at baseline and at various time points during the treatment period, as well as after the completion of the treatment at follow-up 6 months, 1 and 2 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

* IBS diagnosis

Exclusion Criteria:

* Organic GI disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Change in gastrointestinal symptom severity measured by the IBS Severity Scoring System questionnaire (IBS-SSS) | Baseline (week 0), during treatment (week 6), at treatment completion (week 12), follow-up (6 months, 1 and 2 years after treatment initiation)
  The score is calculated from 5 items: pain severity, pain frequency, abdominal bloating severity, bowel habit dissatisfaction and daily life interference. The score ranges from 0-500. A higher the score signifies more severe symptoms. A symptom score reduction of 50 points or more after treatment compared to the baseline score is considered a response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Simrén, Principal Investigator — Göteborg University
Locations (2):
- Sweden (2):
  - Mag-Tarmlab, Sahlgrenska University Hospital, Gothenburg
  - Sahlgrenska University Hospital, Gothenburg

IPD SHARING:
Plan to Share IPD: No